CLINICAL TRIAL: NCT06368882
Title: Efficacy and Safety of Antiviral Therapy With Peg-interferon for Chronic Hepatitis B Complicated With Nonalcoholic Fatty Liver Disease（OCEAN PROJECT）
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yongping _Chen
Record Dates: First submitted 2024-03-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-02

CONDITIONS: Nonalcoholic Fatty Liver Disease; Chronic Hepatitis b
Keywords: Nonalcoholic Fatty Liver Disease; Chronic Hepatitis B; Peg-Interferon α; nucleo(s)tide analogues
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Treatment Group [PEG-IFNα-based antiviral therapy (combined with NAs or PEG-IFNα monotherapy)]: PEG IFNα injection 180 μg is administrated subcutaneously on the first day of the first week, weekly; If HBsAg is negative within 48 weeks of treatment, Peg IFNα combined with NAs or PEG-IFNα monotherapy was continued for 12 weeks, with a maximum of 96 weeks, and the patients are followed up to 240 weeks after the end of treatment. If the patient doesn't achieve HBsAg negative conversion within 48 weeks of treatment, the maximum duration of Peg-IFNα treatment is 96 weeks, and the NAs treatment can be continued until the time of discontinuation where combined treatment programme is used (if HBsAg negative, the consolidation treatment for not less than 24 weeks, and if HBsAg positive still, the treatment with NAs continue). The total of duration of treatment or follow-up is 240 weeks after the end of treatment.
  Interventions: Drug: Peg-Interferon α
- Control Group (No Intervention): Control group (receiving NAs monotherapy) : on the first day of the first week, daily, according to the standard dosage of each drug, until the time when the drug can be stopped (if HBsAg negative conversion is achieved, NAs should be ended after consolidation treatment for not less than 24 weeks; if HBsAg negative conversion is not achieved, NAs therapy should be continued), and follow-up up to 240 weeks after the end of treatment.

INTERVENTIONS:
Drug: Peg-Interferon α — Peg IFN-α injection was subcutaneously injected 180 μg weekly on the first day of the first week, and NAs was administered daily according to the standard dosage of each drug. For example, HBsAg sero-conversion is achieved within 48 weeks of treatment, Peg IFNα combined with NAs or PEG-IFNα monotherapy was continued for 12 weeks, with a maximum of 96 weeks, and follow-up up to 240 weeks after treatment. If HBsAg negative sero-conversion is not achieved within 48 weeks of treatment, the maximum duration of PEG-IFNα is not more than 96 weeks. If Peg IFNα combined NAs regimen is used, NAs can be continued until the drug can be ended (if HBsAg negative conversion is achieved, NAs should be ended after consolidation therapy not less than 24 weeks; if HBsAg negative conversion is not achieved, NAS should be continued), followed up to 240 weeks after treatment.
  Other Names: nucleo(s)tide analogue
  Arms: Treatment Group

SUMMARY:
This is a prospective, multicenter, open-label, non-randomized controlled real-world study to explore the efficacy and safety and to accumulate more evidence-based medical data of an antiviral treatment programme for chronic viral hepatitis B with nonalcoholic fatty liver disease.

A total of 1500 patients with chronic hepatitis B complicated with nonalcoholic fatty liver disease are divided into test group (1000 patients receiving PEG-IFNα-based antiviral therapy (combined NAs or Peg-IFNα monotherapy) and control group（500 patients receiving NAs monotherapy） according to their treatment intention. Laboratory and medical data from specified follow-up points are collected, and adverse events and drug combinations are recorded detailly.

The primary efficacy indicator is HBsAg clearance at 48 weeks of treatment, and the secondary indicators included: (1) HBsAg clearance at 96 weeks of treatment, (2) Cumulative HBsAg clearance at week 24、120、144、168、192、216 and 240; (3) The improvement of liver function level(ALT, AST, TBIL, etc.), blood lipid (TC, TG, LDL-C, HDL-C, etc.), fasting blood glucose, insulin resistance index (HOMA-IR), controlled attenuation parameter, body mass index , liver stiffness measurement, liver histological fibrosis, FIB-4 index from baseline; (4)Incidence of liver cirrhosis and hepatocellular carcinoma during follow-up.

The security assessment includes adverse events, vital signs, and imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-60 years old, male or female (including 18 and 60 years old);
2. meet the diagnostic criteria for chronic hepatitis B in the Guidelines for the prevention and treatment of chronic hepatitis B (2022 edition), and meet the imaging diagnostic criteria for fatty liver in the guidelines for the prevention and treatment of non-alcoholic fatty liver disease (2018 Update edition).
3. serum HBsAg positive >6 months;
4. NAs treatment: baseline HBsAg≤1500 IU/ml, HBeAg negative, HBV DNA negative (not detected);
5. IHC initial treatment: baseline HBsAg<1000 IU/ml, HBeAg negative, HBV DNA negative (undetectable), ALT and AST persistently normal (ULN: <50 IU/L in men, <40 IU/L in women);
6. a negative serum pregnancy test within 24 hours before the first dose (for women of reproductive age);
7. willing to receive treatment and signed informed consent.

Exclusion Criteria:

1. co-infection with active hepatitis A, C, D, E and/or HIV; Or combined with drug-induced liver injury, inherited metabolic liver disease, autoimmune hepatitis, alcoholic liver disease;
2. Liver tumor was detected by liver imaging at the time of screening;
3. patients diagnosed with hepatitis B cirrhosis, that is, those with liver biopsy pathology consistent with liver cirrhosis, or with two or more of the following five criteria, excluding non-cirrhotic portal hypertension: ① imaging examination showed signs of liver cirrhosis and/or portal hypertension; ② Esophagogastric varices were found by endoscopy; ③ Liver stiffness was consistent with cirrhosis; ④ Blood biochemical examination showed decreased albumin level (< 35 g/L) and/or prolonged prothrombin time (prolonged > 3 seconds compared with the control); ⑤ Blood routine examination showed platelet count < 100×109/L;
4. pregnant or lactating women or those who plan to become pregnant and do not want to use contraception during the study period;
5. neutrophil count <1.5×109/L or platelet count <90×109/L. Patients with creatinine higher than 1.5 times the upper limit of normal;
6. The patients and their close relatives (parents, siblings, etc.) had a history of severe mental illness, especially depression. Severe psychosis is defined as severe depression or psychosis, suicide attempt, hospitalization due to psychosis, or a period of incapacitation due to psychosis;
7. patients with a history of immune-mediated diseases (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis) or abnormally elevated levels of autoimmune antibodies;
8. patients with serious diseases of heart, lung, kidney, brain, blood and other important organs, and patients with other malignant tumors;
9. history of severe epilepsy or current use of antiepileptic drugs. Control of unstable diabetes, hypertension, thyroid disease, etc. A history of severe retinopathy or other evidence of retinopathy;
10. any history of organ transplantation and existing functional graft (except corneal or hair transplantation);
11. patients who are allergic to interferon and its drug components, and who are not suitable for interferon according to the investigator's judgment;
12. Patients deemed by the investigator to be ineligible for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance | 48 weeks
  HBsAg clearance at 48 weeks of treatment

SECONDARY OUTCOMES:
HBsAg clearance at 96 weeks | 96 weeks
  HBsAg clearance at 96 weeks of treatment
Cumulative HBsAg clearance rate | week 24、72、120、144、168、192、216、240
  The cumulative clearance rate of HBsAg in chronic hepatitis B patients with different degrees of hepatic steatosis at different treatment nodes; Stratified analysis was performed according to the CAP baseline at enrollment (mild, moderate and severe fatty liver) to explore the correlation between hepatic steatosis and HBsAg clearance rate under different antiviral treatment regimens.
Liver Function Tests | week 24、48、72、96、120、144、168、192、216、240
  the level of ALT and AST
The incidence of liver cirrhosis and liver cancer | week 24、48、72、96、120、144、168、192、216、240
  The incidence of liver cirrhosis and liver cancer

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Ningbo No.2 Hospital, Ningbo
  - Ruian People's Hospital, Rui’an
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou People's Hospital, Wenzhou
  - Yueqing People's Hospital, Yueqing